CLINICAL TRIAL: NCT06062706
Title: Comparison of Outcomes in Robotic vs. Laparoscopic vs. Open Living Donor Hepatectomy: A Single Center Prospective Registry Study
Brief Title: Robotic vs. Laparoscopic vs. Open Living Donor Hepatectomy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: RAC 2121012
Record Dates: First submitted 2023-09-12; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: End Stage Liver Disease; Acute Liver Failure; Acute-On-Chronic Liver Failure; Hepatocellular Carcinoma
MeSH Terms: conditions — End Stage Liver Disease; Liver Failure, Acute; Acute-On-Chronic Liver Failure; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Open: Open donor hepatectomy approach: a portion of the liver is resected from a living donor using the traditional open surgical technique, involving a large incision to access the liver directly. This method is most commonly used in living donor liver transplantation nowadays.
  Interventions: Procedure: Donor hepatectomy
- Laparoscopic: Laparoscopic donor hepatectomy is a minimally invasive surgical approach where a portion of the liver is resected from a living donor using small incisions and specialized instruments.
  Interventions: Procedure: Donor hepatectomy
- Robotic: Robotic donor hepatectomy is an advanced, minimally invasive surgical technique where a portion of the liver is resected from a living donor using robotic instruments. This method is known to provide enhanced precision, improved ergonomics, and superior 3D visualization.
  Interventions: Procedure: Donor hepatectomy

INTERVENTIONS:
Procedure: Donor hepatectomy — Donor hepatectomy is a surgical procedure to resect a portion of the liver from a living donor for transplantation. This usually involved the right lobe, the left lobe or the left lateral section of the liver. Depending on the surgical method, this can be achieved through open, laparoscopic, or robotic-assisted techniques.
  As for the recipient, liver transplantation involves a total hepatectomy of the diseased liver from the recipient and implantation of the liver graft from the donor. This is typically performed using the open surgical approach.
  Other Names: Recipient liver transplantation

SUMMARY:
This will be a study to examine the outcomes of open, laparoscopic, and robotic Living Donor Liver Transplantation (LDLT) procedures. The analysis will encompass 3,448 cases (1,724 donor-recipient pairs) from January 2011 to March 2023, documenting the transition between these surgical techniques, with a noted crossover in 2018.

DETAILED DESCRIPTION:
Background: Liver transplantation is a primary treatment for end-stage liver disease, enhancing survival rates and life quality. Living donor liver transplantation (LDLT) has gained prominence due to the scarcity of deceased donor organs. Historically, the open technique dominated living donor hepatectomies. However, advances in minimally invasive surgery (MIS) led to laparoscopic and later robotic procedures. With the introduction of robotic surgery, MIS for complex surgeries improved, offering better precision and ergonomics.

Objective: To compare the short and long-term outcomes of open, laparoscopic, and robotic LDLT, focusing on both donors and recipients.

Methods: Study Design: Retrospective analysis of data from a prospective liver transplant registry, examining three LDLT techniques.

Setting: King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia.

Participants: All consecutive living donor and recipient pairs undergoing LDLT between January 2011 and March 2023. Exclusions include dual or domino LDLT.

Surgical Techniques: Open, laparoscopic, and robotic techniques used for donor hepatectomies.

Variables: Primary focus on morbidity, conversion rates, and in-hospital mortality for both donors and recipients. Secondary variables will include major complications, graft, and recipient survival rates.

Data Sources and Measurement: Data sourced from a secured, encrypted transplant database, detailing patient data, operation characteristics, and post-op outcomes. Complication severity will be captured using the Clavien-Dindo classification and Comprehensive Complication Index™.

Study Size: Determined by the total number of procedures during the study duration, deemed sufficient for comparison.

Quantitative Variables: Demographics, comorbidities, operational details, post-op and long-term outcomes.

Statistical Methods: Various statistical tests will be employed for comparison, including the Student t, Mann-Whitney U, one-way ANOVA, Fischer and Chi square. Survival will be evaluated using the Kaplan-Meier method. Multivariable binary logistic regression will be employed. All statistical analyses will be conducted using R.

Ethics Approval: Obtained (ID: RAC 2121012) and in accordance with the 1964 Helsinki declaration.

ELIGIBILITY:
Inclusion Criteria:

* All donor and recipient pairs that underwent LDLT at the study institution
* Between 01 January 2011 to 31 March 2023
* Both adult-to-adult and adult-to-pediatric LDLT are included.

Exclusion Criteria:

* Dual and domino LDLT are excluded.

Ages: 1 Month to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study cohort consists of 1,724 living donor and recipient pairs, amounting to a total of 3,448 individuals. These donors and recipients participated in living donor liver transplantation (LDLT) procedures at the King Faisal Specialist Hospital and Research Center in Riyadh, Saudi Arabia.
  The donors provided a portion of their liver for transplantation. The recipient group is diverse, including both adult and pediatric patients receiving transplants from adult donors. Both laparoscopic-assisted and robotic-assisted transplant procedures will be part of the study to ensure an intention-to-treat analysis.
Sampling Method: Non-Probability Sample
Enrollment: 3448 (Estimated)
Dates: Start 2023-08-06 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Donor overall morbidity rate | From date of donor hepatectomy until the date of first hospital discharge assessed up to 90 days postoperatively.
  Complication rate of any severity according to the Clavien-Dindo Classification
Recipient overall morbidity rate | From date of liver transplantation until the date of hospital discharge assessed up to 90 days postoperatively.
  Complication rate of any severity according to the Clavien-Dindo Classification
Recipient in-hospital mortality rate | From date of liver transplantation until the date of death assessed up to 90 days post-transplant.
  Recipient death up to 90 days of follow up

SECONDARY OUTCOMES:
Donor minimally invasive surgery conversion to open rate | Time from operation start until conversion to open in minutes assessed up to 720 min
  Includes conversion to open surgery for both laparoscopic and robotic approaches. This does not apply for the open surgical approach.
Donor hospital stay in days | From date of donor hepatectomy until the date of first hospital discharge assessed up to 90 days postoperatively.
  Number of days the donor was hospitalised during first hospitalisation. Does not include re-hospitalizations.
Recipient Intensive Care Unit (ICU) stay in days | Total number of days hospitalised in ICU, from date of liver transplant until the date of discharge from ICU assessed up to 90 days postoperatively.
  Total number of days recipient stayed in ICU. This included readmissions to ICU.
Recipient hospital stay in days | From date of liver transplant until the date of first hospital discharge assessed up to 90 days postoperatively.
  Number of days the recipient was hospitalised. Does not include rehospitalizations.
Graft survival rates | From date of liver transplantation until the date of re-transplantation or recipient death or last follow up assessed up to 120 months post-transplant
  Graft survival defined as re-transplantation or recipient death.
Recipient survival rates | From date of liver transplantation until the date of recipient death or last follow up assessed up to 120 months post-transplant
  Recipient survival defined as death post-transplant

OTHER OUTCOMES:
Major morbidity rates | From date of operation until the date of hospital discharge assessed up to 90 days postoperatively.
  These include complications of Grade > 2 according to the Clavien-Dindo Classification, i.e., requiring an intervention on the patient requiring organ support in the Intensive Care Unit
Specific complication rates | From date of operation until the date of hospital discharge assessed up to 90 days postoperatively.
  Infection, bleeding, ascites, vascular, and biliary complications

CONTACTS AND LOCATIONS:
Overall Officials: Dieter C Broering, MD, PhD, Principal Investigator — Organ Transplant Center of Excellence, King Faisal Specialist Hospital & Research Centre
Locations (1):
- Organ Transplant Center of Excellence, King Faisal Specialist Hospital & Research Centre, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No